CLINICAL TRIAL: NCT01710410
Title: Pilot Study of Transcranial Direct Current Stimulation (tDCS) as a Smoking Cessation Treatment for Nicotine Dependent Smokers
Brief Title: Transcranial Direct Current Stimulation in a Smoking Cessation Trial
Acronym: tDCS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Nuraleve, Inc. (Industry)
Responsible Party: Principal Investigator, Laurie Zawertailo, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016-2015
Record Dates: First submitted 2012-09-21; First posted 2012-10-19 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Nicotine Dependence
Keywords: transcranial direct current stimulation; nicotine dependence; dorsolateral prefrontal cortex; nicotine replacement therapy; nicotine patch; addiction; smoking cessation; neuroplasticity
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DLPFC tDCS (left anode/right cathode) (Experimental): Active transcranial Direct Current Stimulation (tDCS) administered to the left DLPFC. Brief (20-min) application of weak electric current (e.g., 2 mA) to the scalp.
  Interventions: Device: active transcranial Direct Current Stimulation
- DLPFC tDCS (left cathode/right anode) (Experimental): Active transcranial Direct Current Stimulation (tDCS) administered to the right DLPFC. Brief (20-min) application of weak electric current (e.g., 2 mA) to the scalp.
  Interventions: Device: active transcranial Direct Current Stimulation
- DLPFC tDCS (Sham Comparator): Sham transcranial Direct Current Stimulation (tDCS) delivered to the DLPFC. Brief (30-sec) application of weak electric current (e.g., 2mA) to the scalp.
  Interventions: Device: sham transcranial Direct Current Stimulation

INTERVENTIONS:
Device: active transcranial Direct Current Stimulation — Brief (20-min) application of weak electric current (e.g., 2 mA) to the scalp.
  Arms: DLPFC tDCS (left anode/right cathode); DLPFC tDCS (left cathode/right anode)
Device: sham transcranial Direct Current Stimulation — Brief (30-sec) application of weak electric current (e.g., 2mA) to the scalp.
  Arms: DLPFC tDCS

SUMMARY:
The purpose of this study is to determine the effectiveness of transcranial direct current stimulation (tDCS) plus nicotine patch as a viable smoking cessation program for nicotine dependent smokers.

DETAILED DESCRIPTION:
BACKGROUND: Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation that involves the application of brief weak electric current to the scalp. tDCS may induce neuroplasticity, thereby engaging some of the same systems that figure prominently in the pathological neuroplasticity caused by addictive drugs.

OBJECTIVE: To assess whether tDCS delivered along with nicotine patch reliably increases a) quit rates, b) duration of abstinence, and c) percentage of participants abstinent at follow-up.

METHOD: Active (20min; 2mA) and sham (30sec; 2mA) stimulation will be applied to the dorsolateral prefrontal cortex (DLPFC) in both cerebral hemispheres.

HYPOTHESES:

1. Active tDCS (20-min; 2 mA) will increase abstinence in a standard smoking cessation protocol relative to a sham procedure.
2. The benefits of active left anodal stimulation (anode-left/cathode-right) to the DLPFC will be greater than of active tDCS in the reverse configuration (cathode-left/anode-right).

ELIGIBILITY:
Inclusion Criteria:

* nicotine dependent
* treatment-seeking
* smoke minimum of 15 cigarettes per day
* able to provide written informed consent
* able and willing to attend weekly appointments, inter-treatment and follow-up assessment
* able and willing to wear nicotine patch

Exclusion Criteria:

* currently taking GABA receptor agonists, NMDA receptor antagonists, dopamine receptor agonists/antagonists, SSRIs, L-dopa, anticholinergics
* pregnancy or lactation
* any serious medical condition requiring treatment or medication including high blood pressure, heart problems, asthma, epilepsy
* brain/neurological injury/disease/disorder
* skin disease
* current DSM-IV Axis I psychiatric disorder
* metal or medical device implants
* current treatment for alcohol or drug use
* current use of herbal/holistic preparations
* current use of recreational drugs

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | Participants will be followed for the duration of the study, an expected average of 9 months.
  Measure whether active tDCS increases abstinence in a standard smoking cessation protocol relative to a sham tDCS procedure

OTHER OUTCOMES:
Smoking cessation rate following transcranial direct current stimulation (tDCS) applied to the left dorsolateral prefrontal cortex (DLPFC) versus the right DLPFC. | Participants will be followed for the duration of the study, an expected average of 9 months.
  Measure whether the benefits of active tDCS (anode-left/cathode-right) to the DLPFC will be greater than of active tDCS in the reverse configuration (cathode-left/anode-right) to that region.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Zawertailo, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health (Nicotine Dependence Clinic), Toronto, Ontario, Canada

REFERENCES:
- [Background] Boggio PS, Liguori P, Sultani N, Rezende L, Fecteau S, Fregni F. Cumulative priming effects of cortical stimulation on smoking cue-induced craving. Neurosci Lett. 2009 Sep 29;463(1):82-6. doi: 10.1016/j.neulet.2009.07.041. Epub 2009 Jul 18. PMID 19619607
- [Background] Feil J, Zangen A. Brain stimulation in the study and treatment of addiction. Neurosci Biobehav Rev. 2010 Mar;34(4):559-74. doi: 10.1016/j.neubiorev.2009.11.006. Epub 2009 Nov 13. PMID 19914283
- [Background] Fregni F, Liguori P, Fecteau S, Nitsche MA, Pascual-Leone A, Boggio PS. Cortical stimulation of the prefrontal cortex with transcranial direct current stimulation reduces cue-provoked smoking craving: a randomized, sham-controlled study. J Clin Psychiatry. 2008 Jan;69(1):32-40. doi: 10.4088/jcp.v69n0105. PMID 18312035
- See also: Centre for Addiction and Mental Health (investigator-driven, not initiated, study) — http://www.camh.ca
- See also: Ontario Brain Institute — http://www.braininstitute.ca/
- See also: Nuraleve, Inc. (regulatory sponsor with Health Canada) — http://www.nuraleve.com